CLINICAL TRIAL: NCT04111627
Title: A Feasibility and Pilot Study of Combined Treatment Protocol Using Aerobic Exercise and Duloxetine in Older Adults With Symptomatic Knee Osteoarthritis and Comorbid Depression
Brief Title: Exercise Plus Duloxetine for Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Alan Rathbun, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00089160; K01AG064041 (NIH)
Record Dates: First submitted 2019-09-18; First posted 2019-10-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis; Depression
MeSH Terms: conditions — Osteoarthritis, Knee; Depression | interventions — Exercise; Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aerobic exercise plus Duloxetine (Experimental): Participants will have a starting duloxetine dosage of 30 mg/day and be titrated up to a daily optimal dosage of 60 mg/day as tolerated during the first 12-weeks of the study. Twelve weeks after the receipt of their prescription, participants will be evaluated for the need to increase medication dosage to 90 mg/day. After duloxetine initiation, participants will be provided an exercise prescription that includes a progressive walking program aiming to achieve 50 minutes of moderate-intensity physical activity, three times per week, over 24 weeks.
  Interventions: Behavioral: Aerobic exercise; Drug: Duloxetine

INTERVENTIONS:
Behavioral: Aerobic exercise — Participants with symptomatic knee osteoarthritis and depressive symptoms will be enrolled in a progressive walking program designed to reduce pain and disability and improve psychosocial health.
Drug: Duloxetine — Duloxetine is an FDA-approved selective serotonin and norepinephrine reuptake inhibitor antidepressant approved for the treatment of neuropathic pain in symptomatic knee osteoarthritis as well as depression in adults. Participants with symptomatic knee osteoarthritis and depressive symptoms will receive duloxetine to decrease pain and depression severity to enhance their ability to engage in aerobic exercise.

SUMMARY:
This study evaluates the addition of duloxetine to aerobic exercise in the treatment of symptomatic knee osteoarthritis and depressive symptoms in adults. All participants will receive the receive the treatment protocol, which will first be evaluated in terms of feasibility and then pilot tested.

DETAILED DESCRIPTION:
Symptomatic knee osteoarthritis (OA) affects 10% of men and 13% of women 60 years or older, and depressive symptoms are common, occurring in one-fifth of these patients. Depressive symptoms worsen knee OA disease severity and are a barrier to pain management and engagement in physical activity. Guidelines recommend depression treatment in older adults with knee OA but provide no direction on how to simultaneously manage the co-occurrence of physical and mental morbidity. Treatment recommendations advise exercise to manage pain and disability and improve psychosocial health in knee OA patients; however, compliance to exercise programs is low in persons with chronic pain and disability and is only made worse by comorbid depression. Adherence is critical to the efficacy of depression treatments using exercise training, and no such exercise program has ever been designed for and tested in OA patients with co-occurring depressive symptoms in a way to enhance compliance. Duloxetine is the only antidepressant medication indicated for pain management in knee OA patients that has demonstrated efficacy and tolerability when treating depression in older adults and is a viable pharmacological complement to exercise. There are no protocols that combine treatments using interventions that affect symptoms of both knee OA and depression, and the study goals are to evaluate the feasibility of and then pilot test a protocol comprised of aerobic exercise training plus duloxetine for the treatment of symptomatic knee OA and comorbid depression.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. 40 years or older
3. Symptomatic knee osteoarthritis fulfilling 1986 American College of Rheumatology criteria
4. No plan for surgical knee osteoarthritis intervention within six months of enrollment
5. Major depressive disorder satisfying diagnostic criteria according to the DSM-V
6. Ability to participate in a supervised aerobic exercise program

Exclusion Criteria:

1. Already performing aerobic or resistive exercise 2x/week or more
2. Taking duloxetine, antipsychotics, benzodiazepines, or opioid analgesics
3. Other medications deemed by study team to endanger the health of the participant or unduly confound the results
4. Cognitive impairment (Mini-Mental State Examination score < 20)
5. Past or current bipolar disorder or psychotic symptoms according to the DSM-V
6. Substance abuse disorder or suicidal ideation within the previous year
7. Not able to participate in a supervised exercise program based on the presence of unstable angina, recent MI (within last 3 months), hemiparetic gait, inability to walk at least 1mph on treadmill safely, poorly controlled hypertension (resting blood pressure > 190/110), peripheral arterial disease with current foot or leg ulcers, or cardiac or pulmonary disease with exercise tolerance NYHA class 3 or higher.
8. Active cancer that is currently undergoing treatment (receiving chemotherapy and/or radiation therapy)
9. Pregnant or lactating women
10. Other conditions deemed by study team to endanger the health of the participant or unduly confound the results

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Knee Osteoarthritis Outcomes Scale (KOOS) pain subscale | Change from Baseline Pain Severity at 12 weeks
  The self-reported KOOS pain subscale is sensitive to changes in knee OA symptoms, and consists of nine items scored on a Likert scale (0 [No problems] to 4 [Extreme Problems]) that ranges from 0-36, with higher values indicating greater severity.
Hamilton Depression Rating Scale (HAM-D) | Change from Baseline Depression Severity at 12 weeks
  The HAM-D is clinician-administered, 21-item questionnaire, designed to rate the severity of depression in patients. Individual scores are based on the first 17 items, each with a possible score of 0-4 (0=Absent; 4=Extreme Symptoms) or 0-2 (0=Absent; 2=Frequent), yielding an overall range of 0-54. Higher scores indicate greater depression severity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rathbun AM, Mehta R, Ryan AS, Dong Y, Beamer B, Golden J, Gallo JJ, Luborsky M, Shardell MD, Peer JE, Hochberg MC. Duloxetine plus exercise for knee osteoarthritis and depression: A feasibility study. Osteoarthr Cartil Open. 2023 Dec 8;6(1):100426. doi: 10.1016/j.ocarto.2023.100426. eCollection 2024 Mar. PMID 38130375